CLINICAL TRIAL: NCT06023953
Title: Comparison of Migraine With and Without Aura in a Large Cohort: Characteristics and Response to Remote Electrical Neuromodulation (REN) Treatment
Brief Title: Migraine With and Without Aura Characteristics and Response to Remote Electrical Neuromodulation (REN) Treatment
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE006
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Migraine With Aura; Migraine Without Aura
Keywords: Migraine; Aura; REN; Nerivio
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Migraine with aura (MWA): Patients with migraine who treated their migraine attack with the Nerivio device at least twice and reported having aura in at least two treatment reports
  Interventions: Device: Nerivio device
- Migraine without aura (MWoA ): Patients with migraine who treated their migraine attack with the Nerivio device at least twice and reported the absence of aura in all of their reports, with at least two reports
  Interventions: Device: Nerivio device

INTERVENTIONS:
Device: Nerivio device — REN treatment with Nerivio device

SUMMARY:
This is a Post-marketing, real-world evidence study investigating the safety and efficacy of the acute treatment of migraine with a Remote Electrical Neuromodulation (REN) device (Nerivio) in migraine patients with and without aura, as well as characterizing demographic and attack characteristic differences between migraine patients with and without aura.

Safety will be assessed by the number and type of device-related adverse events. Efficacy will be evaluated as a change in headache pain severity from baseline to 2 hours post-treatment. Disease characteristics will look into demographic and attack differences between patients with and without aura.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, Israel) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients 12 years old and above. It is a wearable device applied to the upper arm.

As part of the sign-up process for the Nerivio app, all patients accept the terms of use which specify that providing personal information is done on their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback. The app includes a secured, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including the presence or absence of aura, pain level (none, mild, moderate, severe), functional disability (none, mild limitation, moderate limitation, severe limitation), presence of associated symptoms (photophobia, phonophobia, and nausea), and an indication of which medications, if any, were taken within that 2-hour time window.

This post-marketing RWE study investigates the safety and efficacy of the Nerivio treatment in patients with and without aura by analyzing data from patients who used the Nerivio device. The following outcomes will be assessed:

1. Migraine clinical characteristics - Headache pain severity, functional disability and presence of associated symptoms at treatment baseline.
2. Consistent efficacy - Pain relief, freedom from pain, functional disability relief, return to normal function (no disability) and freedom from associated symptoms at 2 hours post-treatment relative to baseline in at least 50% of the treatments.
3. Safety - Rate of serious adverse events, and device-related adverse events in the study's period.

Together, these objectives provide a comprehensive evaluation of the effect of REN as a treatment for migraine with or without aura.

ELIGIBILITY:
Inclusion Criteria:

* Users aged 8 years old and above
* Users who treated their migraine attacks with the Nerivio device at least twice
* Users who prospectively reported the presence of aura in at least two treatment reports (reporting at least twice having aura) , OR:
* Users who prospectively reported the absence of aura in all of their reports, with at least two reports

Exclusion Criteria:

* Users who prospectively reported having aura only once

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with migraine by their HCP and were prescribed Nerivio for treatment of acute migraine
Sampling Method: Non-Probability Sample
Enrollment: 31715 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of consistent Headache Relief at 2 Hours Post-treatment between the MWA and MWoA groups | 2 hours
  The difference between the MWA and MWoA groups in the proportion of subjects reporting headache relief at 2 hours post-treatment in at least 50% of all their treatments. Headache relief is defined as an improvement from severe or moderate pain to mild or no pain.
Comparison of Headache Severity at treatment baseline (T=0h) between the MWA and MWoA groups | 0 hours (at baseline)
  The difference between the MWA and MWoA groups in the proportion of subjects reporting severe/moderate headache pain in at least 50% of their attacks.

SECONDARY OUTCOMES:
Comparison of consistent Pain Freedom at 2 Hours Post-treatment between the MWA and MWoA groups | 2 hours
  The difference between the MWA and MWoA groups in the proportion of subjects reporting pain freedom at 2 hours post-treatment in at least 50% of all their treatments. Pain freedom is defined as the disappearance of pain from severe, moderate, or mild at treatment initiation to no pain 2 hours later.
Comparison of Functional Disability at treatment baseline (T=0h) between the MWA and MWoA groups | 0 hours (at baseline)
  The difference between the MWA and MWoA groups in the proportion of subjects reporting severe/moderate disability in at least 50% of their attacks.
Comparison of Photophobia, Phonophobia and Nausea/vomiting presence at treatment baseline (T=0h) between the MWA and MWoA groups | 0 hours (at baseline)
  The difference between the MWA and MWoA groups in the proportion of subjects reporting presence of a specific symptom in at least 50% of their attacks.
Comparison of Consistent Functional Disability Relief at 2 Hours Post-treatment between the MWA and MWoA groups | 2 hours
  The difference between the MWA and MWoA groups in the proportion of subjects reporting functional disability relief at 2 hours post-treatment in at least 50% of all their treatments. Functional disability relief is defined as an improvement of at least one grade from severe, moderate or mild disability from treatment initiation to 2 hours later.
Comparison of Consistent Functional Disability Freedom at 2 Hours Post-treatment between the MWA and MWoA groups | 2 hours
  The difference between the MWA and MWoA groups in the proportion of subjects reporting functional disability freedom at 2 hours post-treatment in at least 50% of all their treatments. Functional disability freedom is defined as the disappearance of disability from severe, moderate, or mild disability at treatment initiation to no disability 2 hours later.
Comparison of Associated Symptoms Freedom at 2 Hours Post-treatment between the MWA and MWoA groups | 2 hours
  The proportion of subjects reporting freedom from each of the migraine-associated symptoms (photophobia, phonophobia, nausea) in at least 50% of their treatments. Associated symptoms freedom is defined as reporting presence of a symptom at treatment initiation and reporting its absence 2 hours later.
Device Related Adverse Events | up to 30 months
  Rate of serious adverse events, and device-related adverse events reported by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, PhD, Principal Investigator — Theranica Bio-Electronics Ltd
Locations (1):
- Theranica Bio-Electronics Ltd, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No